CLINICAL TRIAL: NCT05129124
Title: Insertion Clinical Study to Evaluate the Orientation Characteristics of Multiple Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-012
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (14):
- T01: +6.00 -2.75 x 180 (Experimental): kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
- T02: +6.00-2.75 x 090 (Experimental): kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
- T03: -3.00-2.75 x180 (Experimental): kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
- T04: -3.00 -2.75 x 090 (Experimental): kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
- T05: -9.00 -2.75 x 180 (Experimental): kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
- T06: -9.00 -2.75 x 090 (Experimental): kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
- T07: -12.00 -2.75 x 180 (Experimental): kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
- T08: -12.00-2.75 x 090 (Experimental): kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses
- C01: +6.00 -2.75 x 180 (Active Comparator): Commercially available Ultra for Astigmatism Contact Lenses
  Interventions: Device: Commercially available Ultra for Astigmatism Contact Lenses
- C02: +6.00-2.75 x 090 (Active Comparator): Commercially available Ultra for Astigmatism Contact Lenses
  Interventions: Device: Commercially available Ultra for Astigmatism Contact Lenses
- C03: -3.00-2.75 x180 (Active Comparator): Commercially available Ultra for Astigmatism Contact Lenses
  Interventions: Device: Commercially available Ultra for Astigmatism Contact Lenses
- C04: -3.00 -2.75 x 090 (Active Comparator): Commercially available Ultra for Astigmatism Contact Lenses
  Interventions: Device: Commercially available Ultra for Astigmatism Contact Lenses
- C05: -9.00 -2.75 x 180 (Active Comparator): Commercially available Ultra for Astigmatism Contact Lenses
  Interventions: Device: Commercially available Ultra for Astigmatism Contact Lenses
- C06: -9.00 -2.75 x 090 (Active Comparator): Commercially available Ultra for Astigmatism Contact Lenses
  Interventions: Device: Commercially available Ultra for Astigmatism Contact Lenses

INTERVENTIONS:
Device: kalifilcon A Daily Disposable Toric LD213001 Contact Lenses — kalifilcon A Daily Disposable Toric LD213001 Contact Lenses at different fittings
  Arms: T01: +6.00 -2.75 x 180; T02: +6.00-2.75 x 090; T03: -3.00-2.75 x180; T04: -3.00 -2.75 x 090; T05: -9.00 -2.75 x 180; T06: -9.00 -2.75 x 090; T07: -12.00 -2.75 x 180; T08: -12.00-2.75 x 090
Device: Commercially available Ultra for Astigmatism Contact Lenses — Commercially available Ultra for Astigmatism Contact Lenses at different fittings
  Arms: C01: +6.00 -2.75 x 180; C02: +6.00-2.75 x 090; C03: -3.00-2.75 x180; C04: -3.00 -2.75 x 090; C05: -9.00 -2.75 x 180; C06: -9.00 -2.75 x 090

SUMMARY:
The objective is to evaluate the fit characteristics (primary gaze orientation, rotational recovery, and movement) of kalifilcon A daily disposable toric lenses as compared to commercially available Ultra for Astigmatism lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and have capacity to read, understand and provide written voluntary informed consent.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis.
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent.

Exclusion Criteria:

1. Participating in a conflicting study.
2. Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Schafer, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch and Lomb Site 01, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There are a total of 14 study lens types (8 test contact lenses and 6 comparators contact lenses). Each study lens type will be worn once for approximately 10 minutes.
Units Other Than Participants: Eyes
Groups:
- All Participants Received Kalifilcon LD213001 Contact Lenses & Ultra for Astigmatism Contact Lenses: Participants were given a total of 14 study lens types (8 kalifilcon A Daily Disposable Toric LD213001 Contact Lenses and 6 Commercially available Ultra for Astigmatism Contact Lenses).
  Each study lens type will be worn once for approximately 10 minutes.
Period: Overall Study
Arm/Group | All Participants Received Kalifilcon LD213001 Contact Lenses & Ultra for Astigmatism Contact Lenses
Started | 30; 60 Eyes
Experimental: T01: +6.00 -2.75 x 180 Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses | 30; 60 Eyes
Experimental: T02: +6.00-2.75 x 090 Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses | 30; 60 Eyes
Experimental: T03: -3.00-2.75 x180 Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses | 30; 60 Eyes
Experimental: T04: -3.00 -2.75 x 090 Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses | 30; 60 Eyes
Experimental: T05: -9.00 -2.75 x 180 Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses | 30; 60 Eyes
Experimental: T06: -9.00 -2.75 x 090 Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses | 30; 60 Eyes
Experimental: T07: -12.00 -2.75 x 180 Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses | 30; 60 Eyes
Experimental: T08: -12.00-2.75 x 090 Kalifilcon A Daily Disposable Toric LD213001 Contact Lenses | 30; 60 Eyes
C01: +6.00 -2.75 x 180 Commercially Available Ultra for Astigmatism Contact Lenses | 30; 60 Eyes
C02: +6.00-2.75 x 090 Commercially Available Ultra for Astigmatism Contact Lenses | 30; 60 Eyes
C03: -3.00-2.75 x180 Commercially Available Ultra for Astigmatism Contact Lenses | 30; 60 Eyes
C04: -3.00 -2.75 x 090 Commercially Available Ultra for Astigmatism Contact Lenses | 30; 60 Eyes
C05: -9.00 -2.75 x 180 Commercially Available Ultra for Astigmatism Contact Lenses | 30; 60 Eyes
C06: -9.00 -2.75 x 090 Commercially Available Ultra for Astigmatism Contact Lenses | 30; 60 Eyes
Completed (There are a total of 14 study lens types (8 test contact lenses and 6 comparators contact lenses). Each study lens type will be worn once for approximately 10 minutes.) | 30; 60 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- All Participants Received Kalifilcon LD213001 ContactLenses and Ultra for Astigmatism Contact Lenses: Participants were given a total of 14 study lens types (8 kalifilcon A Daily Disposable Toric LD213001 Contact Lenses and 6 Commercially available Ultra for Astigmatism Contact Lenses).
  Each study lens type will be worn once for approximately 10 minutes.
Arm/Group | All Participants Received Kalifilcon LD213001 ContactLenses and Ultra for Astigmatism Contact Lenses
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.8 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Primary Gaze Orientation at 3 Minutes for the Lenses Inserted at 90 Degrees
Description: Primary gaze orientation is measured in degrees. Measurement Description: Primary gaze is when the patient is looking straight ahead. Orientation refers to how much the contact lens is rotated on the eye. Primary gaze orientation of the contact lens is measured in degrees at the slit-lamp (microscope) using a reticle (protractor). Lens orientation was measured in primary gaze in 5-degree increments. Negative values indicate the contact lens was rotated in the temporal direction. Positive values indicate the contact lens was rotated in the nasal direction. The greater the value (positive or negative) the more the lens is rotated. The absolute value was calculated for all the measurements. The absolute values were used to calculate the mean primary gaze orientation after 3 minutes of contact lens wear. Criteria: P-values ≤0.05 will be considered statistically significant.
Time Frame: 3 minutes
Population: Measurement Description: Lens orientation (in 5-degree increments) was measured in primary gaze (nasal = +, temporal = -)
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Eyes
Arm/Group | All Participants Received Kalifilcon LD213001 ContactLenses and Ultra for Astigmatism Contact Lenses
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 60
degrees
  T01 | 1.3 (3.92)
  C01 | 3.3 (7.47)
  T02 | 2.0 (4.47)
  C02 | 3.0 (9.43)
  T03 | 1.7 (3.79)
  C03 | 4.0 (16.42)
  T04 | 4.2 (13.90)
  C04 | 1.3 (2.60)
  T05 | 3.3 (9.32)
  C05 | 5.3 (9.37)
  T06 | 2.8 (12.78)
  C06 | 5.0 (16.56)
  T07 | 5.7 (11.58)
  T08 | 3.5 (7.09)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 40 days
Arm/Group | All Participants Received Kalifilcon LD213001 ContactLenses and Ultra for Astigmatism Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT05129124/Prot_SAP_000.pdf